CLINICAL TRIAL: NCT03681327
Title: Sleep Infra-slow Oscillations III: an Observational Study in Healthy Subjects and Patients With Sleep Disorders With and Without Closed-loop Stimulation During Sleep
Brief Title: Sleep Infra-slow Oscillations III
Acronym: Sleep-ISO III
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Neurocenter of Southern Switzerland (Other)
Responsible Party: Principal Investigator, Stephany Fulda, Stephany Fulda, Principal Investigator, Neurocenter of Southern Switzerland
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: EOC.NSI.LS.18.1
Record Dates: First submitted 2018-09-20; First posted 2018-09-24 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sensory stimulation during sleep — Sensory stimulation during sleep

SUMMARY:
In young healthy subjects, we will apply sensory stimuli at specific times during sleep to evaluate the probability that the stimulus evokes an arousal.

ELIGIBILITY:
Inclusion Criteria:

* Willingness to participate and written informed consent
* Aged 20 to 40 years at the time of screening
* Body mass index (BMI) ≤ 30

Exclusion Criteria:

* Pregnancy or breast feeding at the time of screening
* Sleep related breathing disorders
* Any other sleep related breathing disorder according to AASM criteria
* Current history of psychiatric disorders according to DSM-V
* Current chronic treatment that may affect sleep
* Any significant neurological disorder or other medical disease that may affect sleep
* Any unstable medical condition
* Any clinically significant sleep disorder

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 17 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

PRIMARY OUTCOMES:
Arousal probability | 8 hours
  Number stimuli that are followed by an EEG arousal divided by the total number of stimuli

CONTACTS AND LOCATIONS:
Overall Officials: Stephany Fulda, PhD, Principal Investigator — Neurocenter of Southern Switzerland
Locations (1):
- Neurocenter of Southern Switzerland, Lugano, Canton Ticino, Switzerland

IPD SHARING:
Plan to Share IPD: Yes
The data and metadata generating in this project will be deposited onto existing public repositories.